CLINICAL TRIAL: NCT03882203
Title: Cladribine With Intermediate Cytarabine, G-CSF and VP16 Sequential With Fludarabine and Busulifan as Condoning Regimen for Refractory Acute Leukemia
Brief Title: CLAGE Sequential With Flu-Bu Conditioning for Refractory Acute Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, Blood & Marrow Transplantation program, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJH-Ref-AL-2018
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Refractory Hematologic Cancer; Allogeneic Stem Cell Transplantation
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): Patients receive the study protocol: CLAGE sequential with Flu-Bu as conditioning regimen followed by low-dose decitabine maintenance
  Interventions: Drug: CLAGE-FluBu

INTERVENTIONS:
Drug: CLAGE-FluBu — Cladribine combined with cytarabine and VP16 sequential with Fludarabine combined with busulifan

SUMMARY:
For patients with refractory acute leukemia, allogeneic stem cell transplantation is the only curative therapy. Only 20% of patients may achieve long-term survival mostly due to relapse or nor-relapse mortality (NRM). In previous study, we demonstrated that intensive leukemia debulking chemotherapy FLAG-IDA sequential with Flu-BU conditioning is feasible with ~40% long-term survival. In the study, we further modified the chemotherapy with cladribine replacing fludarabine aiming a more potent anti-leukemia effect. Meanwhile, we reduce the dose of busulfan for patients with poor performance status and age over 45 aim to reduce the NRM. All patients will also receive post-transplantation maintenance therapy with low-dose decitabine to prevent relapse.

DETAILED DESCRIPTION:
For patients with refractory acute leukemia, allogeneic stem cell transplantation is the only curative therapy. Only 20% of patients may achieve long-term survival mostly due to relapse or nor-relapse mortality (NRM). In previous study, we demonstrated that intensive leukemia debulking chemotherapy FLAG-IDA sequential with Flu-BU conditioning is feasible with ~40% long-term survival. The most important cause of treatment failures were relapse and non-relpase mortality. The further analysis demonstrated that patients with higher bone marrow blast before allo-HSCT was associated with treatment failure and patients with poor perforce status or age over 45 had increased rate of NRM. To further optimization the protocol, we modified the chemotherapy with cladribine replacing fludarabine aiming a more potent anti-leukemia effect and replace idarubicin with VP-16. All patients will also receive post-transplantation maintenance therapy with low-dose decitabine (5mg/m2 daily for 5 days) to prevent the further reduce the relapse incidence. We anticipate LFS at 1 year should be above 50% and 1-year LFS of 20% is considered unacceptable.

ELIGIBILITY:
Inclusion Criteria:

* refractory myeloid malignancies including acute myeloid leukemia (AML) or chronic myeloid leukemia in blastic crisis (CML-BC)
* HLA matched sibling，unrelated donor, or haplo-identical donor
* Patients with bone marrow blast >5% and positive measurable disease via flowcytometry or PCR.

Exclusion Criteria:

* patients with active infection
* liver function damage: ALT/AST above 2X normal range; and renal function damage Scr>160µmol/L; insufficient pulmonary function (FEV1，FVC，DLCO<50%）and heart failure or with EF <50%
* mental instability
* unwilling to give inform consent

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
leukemia-free survival | 1 year
  From enrollment to any event as relapse or death

SECONDARY OUTCOMES:
overall survival | 1 year
  From enrollment to death
relapse rate | 1 year
  From enrollment to documentation of relapse
non relapse mortality | 1 year
  From enrollment to documentation of death without evidence of leukemia

CONTACTS AND LOCATIONS:
Overall Officials: Junming Li, M.D, Study Director — Department of Hematology, Rui Jin Hospital
Locations (1):
- Blood & Marrow Transplantation Center, RuiJin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No